CLINICAL TRIAL: NCT04103892
Title: A Two-Part Study of CLE-100 as an Adjunct Therapy in Subjects With Major Depressive Disorder
Brief Title: A Study of CLE-100 (Oral Esketamine) in Addition to Standard Antidepressant Drug for Major Depressive Disorder - CLEO Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Clexio Biosciences Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLE100-MDD-201
Record Dates: First submitted 2019-09-09; First posted 2019-09-26 (Actual); Results first posted 2025-09-24 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-09

CONDITIONS: Adjunctive Treatment of Major Depressive Disorder
Keywords: MDD; depression; depressive disorder; major depression; adjunct therapy; oral; esketamine
MeSH Terms: conditions — Depression; Depressive Disorder; Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: Part A - 16 patients, 2 arms, parallel; Part B - 130 patients, 2 arms, parallel
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part A - CLE-100 (oral esketamine) (Experimental): Part A: 1 oral tablet of CLE-100 once daily for 1 week.
  Interventions: Drug: CLE-100
- Part A - Placebo (Placebo Comparator): Part A: 1 oral tablet of Placebo once daily for 1 week.
  Interventions: Drug: placebo
- Part B - CLE-100 (oral esketamine) (Experimental): Part B: 1 oral tablet of CLE-100 once daily for 4 weeks.
  Interventions: Drug: CLE-100
- Part B - Placebo (Placebo Comparator): Part B: 1 oral tablet of Placebo once daily for 4 weeks.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: CLE-100 — 1 tablet of CLE-100 administered once daily
  Arms: Part A - CLE-100 (oral esketamine); Part B - CLE-100 (oral esketamine)
Drug: placebo — 1 tablet of placebo administered once daily
  Arms: Part A - Placebo; Part B - Placebo

SUMMARY:
The clinical trial is a Phase 2, double-blind, randomized, placebo controlled study in Major Depressive Disorder (MDD) participants currently treated with antidepressant therapy. The objective of the study is to assess CLE-100 for the treatment of MDD in participants currently treated with standard antidepressant therapy.

DETAILED DESCRIPTION:
CLEO study is performed in two parts (part A and Part B). Part A will be an inpatient study to assess the safety, tolerability, and pharmacokinetics of CLE-100 (oral esketamine) in MDD participants currently treated with an antidepressant drug. It will include a screening phase (up to 35 days), a 1 week inpatient double-blind treatment phase and an outpatient post treatment safety follow-up phase of 1 week after last study drug administration.

Part B will be a study to assess the safety and efficacy of CLE-100 (oral esketamine) in MDD participants currently treated with an antidepressant drug with inadequate response to standard antidepressant therapy.

The participants will remain on their current antidepressant therapy with no dose change during the study.

ELIGIBILITY:
Part A - Inclusion Criteria:

1. Male or female between 18 to 60 years of age
2. Primary diagnosis of MDD, without psychotic features according to DSM-5 and supported by the Mini International Neuropsychiatric Interview (MINI)
3. MADRS score of at least 18 at Screening
4. Treatment with stable dose of the current antidepressant therapy for at least 4 weeks for the current major depressive episode (MDE)
5. Body mass index (BMI) between 18 and 40 kg/m2, inclusive
6. Is able and competent to read and sign the informed consent form (ICF).

Part A - Exclusion Criteria:

1. History of substance use disorder per DSM-5 criteria, except for tobacco use disorder
2. History or current diagnosis of bipolar disorder, schizophrenia, schizoaffective disorders, binge eating disorder dementia, delirium, amnesia, or any other significant cognitive disorder
3. Posttraumatic stress disorder, obsessive compulsive disorder, or any other mental disorder (including personality disorders)
4. Has any medical condition for which an increase in blood pressure or intracranial pressure poses a serious risk
5. Female of childbearing potential without appropriate contraceptive means, pregnant or breastfeeding

Part B - Inclusion Criteria:

1. Male or female between 18 to 65 years of age
2. Primary diagnosis of MDD without psychotic features according to DSM-5 and supported by the Mini International Neuropsychiatric Interview (MINI)
3. MADRS score of at least 24 at Screening.
4. At least 2 inadequate responses to antidepressant therapy (ADT) in the current Major Depressive Episode (MDE)
5. Current MDE for at least 12 weeks
6. BMI between 18 and 40 kg/m2, inclusive.
7. Is able and competent to read and sign the ICF.

Part B - Exclusion Criteria:

1. Inadequate response to more than 5 treatment courses of antidepressant medication therapy during the current MDE
2. Current MDE for longer than 5 years.
3. 3. Has a current substance use disorder or history of any substance use disorder per DSM-5 criteria within 12 months prior to Screening, except for tobacco use disorder.
4. Has a history or current diagnosis of bipolar disorder, schizophrenia, or schizoaffective disorders.
5. Has dementia, delirium, amnesia, or any other significant cognitive disorder.
6. Has posttraumatic stress disorder, obsessive compulsive disorder, or any other mental disorder (including personality disorders, eating disorders, etc.).
7. Has any medical condition for which an increase in blood pressure or intracranial pressure poses a serious risk.
8. Has been randomized in Part A of this study.
9. Is a female of childbearing potential pregnant or breastfeeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2019-09-05 (Actual); Primary Completion 2022-09-21 (Actual); Study Completion 2022-10-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (46):
- United States (45):
  - Clinical Site 126, Bentonville, Arkansas
  - Clinical Site 120, Little Rock, Arkansas
  - Clinical Site 129, Little Rock, Arkansas
  - Clinical Site 141, Anaheim, California
  - Clinical Site 115, Bellflower, California
  - Clinical Site 132, Lafayette, California
  - Clinical Site 117, Oakland, California
  - Clinical Site 113, Oceanside, California
  - Clinical Site 123, Riverside, California
  - Clinical Site 124, Santa Ana, California
  - Clinical Site 142, Santa Rosa, California
  - Clinical Site 112, Torrance, California
  - Clinical Site 145, Denver, Colorado
  - Clinical Site 107, Hialeah, Florida
  - Clinical Site 116, Miami, Florida
  - Clinical Site 108, Miami Gardens, Florida
  - Clinical Site 105, Orlando, Florida
  - Clinical Site 137, Orlando, Florida
  - Clinical Site 140, Atlanta, Georgia
  - Clinical Site 104, Decatur, Georgia
  - Clinical Site 122, Marietta, Georgia
  - Clinical Site 131, Baltimore, Maryland
  - Clinical Site 136, Rockville, Maryland
  - Clinical Site 103, Boston, Massachusetts
  - Clinical Site 121, Boston, Massachusetts
  - Clinical Site 151, Dearborn Heights, Michigan
  - Clinical Site 139, St Louis, Missouri
  - Clinical Site 125, Lincoln, Nebraska
  - Clinical Site 110, Las Vegas, Nevada
  - Clinical Site 101, Marlton, New Jersey
  - Clinical Site 148, Toms River, New Jersey
  - Clinical Site 128, New York, New York
  - Clinical Site 102, Staten Island, New York
  - Clinical Site 111, Hickory, North Carolina
  - Clinical Site 143, Raleigh, North Carolina
  - Clinical Site 138, Middleburg Heights, Ohio
  - Clinical Site 127, North Canton, Ohio
  - Clinical Site 106, Media, Pennsylvania
  - Clinical Site 118, Philadelphia, Pennsylvania
  - Clinical Site 114, Fort Worth, Texas
  - Clinical Site 109, Houston, Texas
  - Clinical Site 149, Missouri City, Texas
  - Clinical Site 144, Plano, Texas
  - Clinical Site 147, Draper, Utah
  - Clinical Site 135, Bellevue, Washington
- Clinical Site 150, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Part A - CLE-100 (Oral Esketamine) | Part A - Placebo | Part B - CLE-100 (Oral Esketamine) | Part B - Placebo
Started | 13 | 3 | 72 | 58
Completed | 12 | 3 | 66 | 48
Not Completed | 1 | 0 | 6 | 10
Not completed — Adverse Event | 0 | 0 | 0 | 3
Not completed — Lost to Follow-up | 0 | 0 | 2 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 2 | 5
Not completed — Requirement of prohibited concomitant medication | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A - CLE-100 (Oral Esketamine) | Part A - Placebo | Part B - CLE-100 (Oral Esketamine) | Part B - Placebo | Total
Number analyzed (Participants) | 13 | 3 | 72 | 58 | 146
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.23 (9.99) | 49.00 (7.55) | 42.79 (13.24) | 46.19 (13.14) | 44.93 (12.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 51 | 43 | 101
  Male | 8 | 1 | 21 | 15 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 15 | 24 | 40
  Not Hispanic or Latino | 11 | 3 | 57 | 33 | 104
  Unknown or Not Reported | 1 | 0 | 0 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 6 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 10 | 3 | 11 | 10 | 34
  White | 3 | 0 | 54 | 46 | 103
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  Puerto Rico | 0 | 0 | 2 | 0 | 2
  United States | 13 | 3 | 70 | 58 | 144

OUTCOME MEASURES:

1. Primary Outcome: Part B - Change From Baseline in Montgomery-Asberg Depression Rating Scale (MADRS) Score
Description: The MADRS is a validated clinician-administered measurement of depression severity commonly used in clinical trials of depression treatments to select subjects and assess efficacy. The test consists of 10 items, each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total possible score of 60. Higher scores represent a more severe condition.
Time Frame: 29 days
Population: The Full Analysis Set (FAS), which is a subset of the ITT Analysis Set, includes all data collected while on study drug for all randomized subjects who received at least 1 dose of study drug during Part B and have both Baseline and at least 1 post-baseline MADRS total score. This Analysis Set serves as the principal analysis set for inference.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Part B - CLE-100 (Oral Esketamine) | Part B - Placebo
Number analyzed (Participants) | 70 | 55
units on a scale | -10.72 (1.13) | -9.46 (1.31)
Statistical Analysis 1: Comparison: Part B - CLE-100 (Oral Esketamine) vs Part B - Placebo; Test type: Superiority; p = 0.46, Mixed Models Repeated Measures (MMRM; Least square (LS) mean difference = -1.26, 95% CI 2-sided [-4.60 to 2.09], Standard Error of Mean 1.69

2. Post Hoc Outcome: Part B - Change From Baseline in Montgomery-Asberg Depression Rating Scale (MADRS) Score in 2022 Cohort (Corresponding to a Post-acute Phase of the COVID-19 Pandemic)
Description: as for outcome 1
Time Frame: 29 days
Population: 2022 cohort (corresponding to a post-acute phase of the COVID-19 pandemic) of the Full Analysis Set (FAS) includes all data collected while on study drug for all randomized subjects in 2022 who received at least 1 dose of study drug during Part B and have both Baseline and at least 1 post-baseline MADRS total score. This Analysis Set serves as the principal analysis set for inference.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Part B - CLE-100 (Oral Esketamine) | Part B - Placebo
Number analyzed (Participants) | 35 | 30
units on a scale | -12.96 (1.60) | -7.68 (1.84)
Statistical Analysis 1: Comparison: Part B - CLE-100 (Oral Esketamine) vs Part B - Placebo; Test type: Superiority; p = 0.03, Mixed Models Repeated Measures (MMRM); Least square (LS) mean difference = -5.28, 95% CI 2-sided [-9.91 to -0.65], Standard Error of Mean 2.34

ADVERSE EVENTS:
Time Frame: Part A: 2 weeks; Part B: 6 weeks
Arm/Group | Part A - CLE-100 (Oral Esketamine) | Part A - Placebo | Part B - CLE-100 (Oral Esketamine) | Part B - Placebo
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/3 | 0/72 | 0/57
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/3 | 0/72 | 0/57
Other Adverse Events (participants affected / at risk) | 6/13 | 1/3 | 37/72 | 23/57
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A - CLE-100 (Oral Esketamine) (N=13) | Part A - Placebo (N=3) | Part B - CLE-100 (Oral Esketamine) (N=72) | Part B - Placebo (N=57)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 6 (10) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Feeling abnormal (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood pressure diastolic increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urine analysis abnormal (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Blood pressure systolic increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 9 (11) | 5 (5)
Dizziness (Nervous system disorders) | 4 (4) | 0 (0) | 10 (17) | 1 (2)
Somnolence (Nervous system disorders) | 2 (2) | 0 (0) | 8 (9) | 1 (1)
Sedation (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (6) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypersomnia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypogeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Dissociation (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (3)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Abnormal dreams (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Anger (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bradyphrenia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enuresis (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Euphoric mood (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After the multicenter publication or 18 months after completion of the Study, whichever occurs first, Institution may itself publish the results of its data from the Study. Institution and Principal Investigator shall provide Sponsor with an advance copy of any proposed publication or oral presentation at least 60 days prior to the planned date of submission or presentation and Sponsor shall have 60 days to review the proposed publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-03): https://cdn.clinicaltrials.gov/large-docs/92/NCT04103892/Prot_SAP_000.pdf